CLINICAL TRIAL: NCT02515513
Title: The Role of Muscle Cachexia in Pancreatic Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Original PI left the institution. No subjects enrolled
Sponsor: University of Florida (Other)
Collaborators: The V Foundation for Cancer Research (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201500239 - N; 2R01AR060209-06A1 (NIH)
Record Dates: First submitted 2015-06-03; First posted 2015-08-04 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Pancreas Cancer
Keywords: Pancreas; Pancreas Cancer; Muscle Biopsy; Cachexia; Muscle Cachexia
MeSH Terms: conditions — Pancreatic Neoplasms; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pancreatic Cancer Patients (Active Comparator): During the surgical resection for the pancreatic cancer a muscle tissue biopsy sample will be performed.
  Interventions: Procedure: Muscle Tissue Biopsy Sample
- Surgical Patients with benign pathology (Active Comparator): During surgical resection for patients with benign right upper quadrant pathology, a muscle tissue biopsy sample will be performed.
  Interventions: Procedure: Muscle Tissue Biopsy Sample

INTERVENTIONS:
Procedure: Muscle Tissue Biopsy Sample — During surgical resection, to enter the abdominal cavity, anterior muscle groups such as the rectus abdominous muscle. This group of muscle is divided. During division, muscle fibers are released from fascial group and discarded off the operative field. This will be the target for specimen collection.

SUMMARY:
The relationship between myopenia, nutritional status, and long-term oncologic outcomes remains poorly characterized in patients with anatomically resectable pancreatic cancer (PC). The investigators want to look at muscle properties in pancreatic cancer patients to determine possible therapeutic options toward better nutritional status. Patients with benign right upper quadrant pathology will be utilized as controls for the study.

The researchers hypothesize that improving cancer cachexia in PC will improve the quality of life and ultimately increase overall survival. The long term goal of is to identify areas of intervention to prevent and/or improve cachectic events in PC in order to significantly improve clinical outcomes. The first step in this long term goal is to fully characterize cachexia in the condition of PC. This research is to understand and modify the local response within skeletal muscle leading to a clinically relevant persistent wasting and to understand and interrupt the systemic stimulus produced by the tumor local environment resulting in these muscle specific mechanisms.

DETAILED DESCRIPTION:
Cancer cachexia (CC) is a devastating condition affecting up to 80% of cancer patients, diminishing quality of life and contributing to increased mortality. Cancer cachexia is a complex metabolic syndrome characterized by the loss of skeletal muscle mass and weakness. The muscle pathology of cancer cachexia is not only related to muscle atrophy but also to disruptions to the contractile apparatus of the muscle. While physiologic disruptions in muscle sarcomere and myofiber membrane integrity have been observed despite the lack of injury, the totality of the muscle specific mechanisms contributing to these phenotypes have not been described, nor investigated in the context of pancreatic cancer (PC) where cachexia is a significant clinical problem. Therefore, delineating specific mechanisms of muscle catabolism in PC is critical to developing clinical therapies to control wasting and improve patient quality of life, clinical outcomes and long-term survival.

A variety of tumor promoting and inflammatory cell signaling pathways have been implicated in cancer cachexia, whereby pro-inflammatory cytokines have been implicated as a driving force. Remarkably, approximately half of all patients with PC demonstrate a measurable acute phase response, which is associated with poor clinical outcomes. Importantly, systemic elevations of these inflammatory mediators are due to a complex local interplay between the developing tumor and the immune system which subsequently leads to a systemic chronic inflammatory state. PC appears to manipulate the immune system to promote its survival at the expense of nutritional stores which results in cachexia. Therefore, understanding of the local and systemic inflammatory response in PC and its relation to muscle specific mechanisms is crucial to developing effective therapies for cancer cachexia.

PC associated cachexia results in a significant therapeutic dilemma. Local approaches such as surgery for curative intent encounter a high recurrence rate which is indicative of the systemic nature of even very early-stage disease. Therefore, systemic therapies are necessary for long-term survival. Unfortunately, effective chemotherapies are only offered to patients with good clinical parameters such as nutritional status. In other words, if the patient is too weak, they are not offered effective therapies for the risk of causing more harm than good.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic Cancer Patients who are potentially surgically resectable.

Exclusion Criteria:

* Patients who do not meet the criteria for surgical resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Ultrastructural abnormalities in muscle tissue samples between the groups | day 1
  To look at the extent of ultrastructural abnormalities in the skeletal muscle by histologic examination of muscle biopsies
Myofiber atrophy in muscle tissue samples between the groups | day 1
  2) identify the growth and atrophy-related transcription factors associated with the muscle pathology and 3) identify the genome-wide gene networks and biological process associated with skeletal muscle pathology in surgically resected PC patients and healthy control patients by RT-PCR and histologic staining of tissues for transcriptional factors associated with cachexia.
Identify gene networks within the skeletal muscle between the groups | day 1
  RT-PCR of RNA from biopsied muscle tissues

SECONDARY OUTCOMES:
History of weight lost | Baseline
  Clinical assessment at treatment follow-up
Nutritional status | Approximately 2 years
  Clinical assessment at treatment follow-up
Blood Chemistry composite | Approximately 2 years
  Clinical assessment at treatment follow-up
Preoperative sarcopenia using a muscular index | Approximately 2 years
  Clinical assessment at treatment follow-up and radiographic measurements of muscle groups on routine surveillance for cancer recurrence or advancement
Measurement of lymphatic metastasis | Approximately 2 years
  Pathologic specimen at time of resection to determine extent of pathologic stage which is routine
Tumor grade | Approximately 2 years
  Noted at pathologic assessment and part of routine examination
Survival data | Approximately 2 years
  Noted on routine follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Judge, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

REFERENCES:
- [Background] Tisdale MJ. Mechanisms of cancer cachexia. Physiol Rev. 2009 Apr;89(2):381-410. doi: 10.1152/physrev.00016.2008. PMID 19342610
- [Background] Evans WJ, Morley JE, Argiles J, Bales C, Baracos V, Guttridge D, Jatoi A, Kalantar-Zadeh K, Lochs H, Mantovani G, Marks D, Mitch WE, Muscaritoli M, Najand A, Ponikowski P, Rossi Fanelli F, Schambelan M, Schols A, Schuster M, Thomas D, Wolfe R, Anker SD. Cachexia: a new definition. Clin Nutr. 2008 Dec;27(6):793-9. doi: 10.1016/j.clnu.2008.06.013. Epub 2008 Aug 21. PMID 18718696